CLINICAL TRIAL: NCT01477359
Title: Cardiac Sarcoidosis Multi-Center Prospective Cohort Study
Brief Title: Cardiac Sarcoidosis Multi-Center Prospective Cohort
Acronym: CHASM-CS
Status: Recruiting | Type: Observational
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: UOHI-04
Record Dates: First submitted 2011-11-10; First posted 2011-11-22 (Estimated); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Cardiac Sarcoidosis
Keywords: Sarcoidosis
MeSH Terms: conditions — Sarcoidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Frozen plasma, serum and buffy coat.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CS screened as underlying etiology: 1. Patients with active Clinically Manifest CS
  2. Patients diagnosed with extra-cardiac sarcoidosis and being screened for CS

SUMMARY:
Recent data has shown that sarcoidosis, presenting initially with cardiac manifestations (CS) of either conduction system disease or cardiomyopathy and sustained VT, is not uncommon. A Canadian physician survey found that most physicians do not investigate for CS as a possibility in these situations. Thus many patients with clinically important CS are going un-diagnosed. A study from Finland showed that missing the diagnosis of CS in these patients' leads to significant mortality and morbidity.

There are no published clinical consensus guidelines on treatment of CS. Corticosteroid therapy is advocated by most experts. This is based on very modest data from small retrospective observational studies using variable definitions of clinical response. The effect of corticosteroid treatment on the clinical course of CS has not been studied in prospective studies and will be one of the aims of this project. Recent physician surveys regarding CS, in Canada and the US, found that current clinical practice varies widely. The 2008 American College of Cardiology/American Heart Association/Heart Rhythm society guidelines recommend implantation of a defibrillator (Class IIa recommendation) to prevent sudden cardiac death. The most recent Canadian device therapy guidelines do not mention CS.

A multi-center collaborative approach to study CS is greatly needed." The investigators propose exactly that i.e. a multi-center prospective cohort to start to answer clinical questions. The investigators have formed the CANADIAN CARDIAC SARCOIDOSIS RESEARCH GROUP. The group includes respirologists with an interest in sarcoidosis, cardiac electrophysiologists, cardiac imaging specialists with extensive experience in imaging of sarcoidosis and biostatisticians. The research will be in two phases; a registry of current diagnostic approaches, treatment and prognosis, and a randomized clinical trial of the effect of corticosteroid treatment on the clinical course of cardiac sarcoidosis.

DETAILED DESCRIPTION:
Baseline assessment of Clinically Manifest CS patients consists of: history, echocardiogram, ECG, chest CT scan, FDG-PET scan, blood for biomarkers within 2 months of the PET scan, cardiac MRI and possibly a signal average ECG and biopsy (encouraged-either endomyocardial or extra-cardiac).

Follow-up and clinical management of clinically manifest patients diagnosed with CS will occur at 3-6 months with a repeat FDG-PET scan and blood biomarkers. Follow-up will then be annually with an echo and ECG. Treatment with steroids/immunosuppressants and device therapy will be at the discretion of the treating physician.

Baseline assessment of patients diagnosed with extra-cardiac sarcoidosis and being screened for CS consists of: history, echocardiogram, ECG, holter, chest CT scan, biopsy, and cardiac MRI (CMR). If the CMR is suggestive of CS the patient will be have a FDG-PET scan done and be followed as a Clinically Silent patient. They will be contacted every 2 years. If the CMR is negative the patient will be followed as a extra-cardiac sarcoidosis patient with no evidence of CS and be in the control group. They will be contacted at 5 years and at the time of study completion.

All patients will be followed until the last patient recruited has been followed for 4 years.

The occurrence of the primary and secondary outcomes will be assessed in treated and untreated patients.

There will be 2 imaging core labs. The PET core lab will be located at UOHI under the direction of Dr. Robert Beanlands. The CMR core lab will be under the direction of Dr. Mathias Friedrich (McGill University). All scans will be read in the core labs by physicians who are blinded to the clinical details of the patients.

The Biomarker core lab will be at The University of Ottawa Heart Institute under the leadership of Dr P Liu.

ELIGIBILITY:
Inclusion Criteria:

To diagnose Clinically Manifest CS all following criteria must be met:

(i) Positive biopsy* for Sarcoid (either EMB or extra-cardiac) AND/OR (ii) CT Chest highly suggestive of pulmonary sarcoidosis AND (iii) one or more of the following clinical features:

* advanced conduction system disease (sustained Mobitz II AV block or third degree AV block)
* non- sustained or sustained ventricular arrhythmia
* ventricular dysfunction (LVEF < 50% and/or RVEF < 40%) AND (iv) No alternative explanation for clinical features AND (v) FDG-PET suggestive of active CS

To diagnose clinically silent CS all of the following criteria must be met

(i) Biopsy proven extra-cardiac sarcoidosis

AND/OR (ii) CT Chest highly suggestive of pulmonary sarcoidosis

AND (iii) CMR suggestive of cardiac sarcoidosis

AND (iv) Does not have criteria for clinically manifest CS ie. should not have any of following

* advanced conduction system disease (sustained Mobitz II AV block or third degree AV block)
* non- sustained or sustained ventricular arrhythmia
* ventricular dysfunction (LVEF < 50% and/or RVEF < 40%)

Patients with negative CMR will be designated as 'extra-cardiac sarcoidosis with no evidence of CS' and followed as control

Exclusion Criteria:

* unable or unwilling to provide informed consent
* patients who are pregnant or lactating
* patients with known claustrophobia
* age < 18 years

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Electrophysiology Service patients
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2012-08; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Clinically Manifest Patients | On active therapy for 6 months
  "Clinically improved" if they are alive and not had a heart transplant and have not had heart failure hospitalization and no sustained VT/VF and meet one or more of following
  (i) No sustained VT (if presented with sustained VT) (ii) Improvement in LV function (defined as 10% decrease in LV end systolic volume or 5% absolute increase in LVEF) (iii) Resolution of conduction system disease (if presented with sustained heart block)
  failure hospitalization and have not had sustained VT and one or both of: a. LV function improvement (defined as 10% decrease in LV end systolic volume) b. Resolution of conduction system disease.
Clinically Silent and Control Patients | 9 years
  Cardiac death or cardiac transplantation or sustained VT/VF or sustained second or third degree AV block or development of clinical congestive heart failure (with documented LVEF < 50%).

SECONDARY OUTCOMES:
total mortality | 6 months and 60 months
cardiovascular mortality | 6 months and 60 months
heart failure hospitalization | 6 months and 60 months
change in LVEF from baseline | 6 months and 60 months
change in disease activity as assessed by PET imaging | 6 months and 60 months
  comparing pre-treatment to 6 month scans
Atrial Fibrillation burden | 6 months and 60 months
  from defibrillator diagnostics
Ventricular arrhythmia burden | 6 months and 60 months
  from defibrillator diagnostics
% of ventricular pacing | 6 months and 60 months

CONTACTS AND LOCATIONS:
Overall Officials: David Birnie, MD, Principal Investigator — Ottawa Heart Institute Research Corporation; Pablo Nery, MD, Principal Investigator — Ottawa Heart Institute Research Corporation; Rob Beanlands, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (14):
- Canada (13):
  - Libin Cardiovascular Institute of Alberta, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - St. Paul's Hospital, Vancouver, British Columbia
  - QEII Health Sciences Center, Halifax, Nova Scotia
  - Hamilton Health Sciences Centre, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Centre Hospitalier de l"Universite de Montreal-Hotel Dieu, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Prairie Vascular Research Inc-Regina General Hospital, Regina, Saskatchewan
- Hokkaido University, Sapporo, Japan

REFERENCES:
- [Derived] Weng W, Wiefels C, Chakrabarti S, Nery PB, Celiker-Guler E, Healey JS, Hruczkowski TW, Quinn FR, Promislow S, Medor MC, Spence S, Odabashian R, Alqarawi W, Juneau D, de Kemp R, Leung E, Beanlands R, Birnie D. Atrial Arrhythmias in Clinically Manifest Cardiac Sarcoidosis: Incidence, Burden, Predictors, and Outcomes. J Am Heart Assoc. 2020 Sep;9(17):e017086. doi: 10.1161/JAHA.120.017086. Epub 2020 Aug 20. PMID 32814465
- [Derived] Martineau P, Pelletier-Galarneau M, Juneau D, Leung E, Nery PB, de Kemp R, Beanlands R, Birnie D. Imaging Cardiac Sarcoidosis With FLT-PET Compared With FDG/Perfusion-PET: A Prospective Pilot Study. JACC Cardiovasc Imaging. 2019 Nov;12(11 Pt 1):2280-2281. doi: 10.1016/j.jcmg.2019.06.020. Epub 2019 Aug 14. No abstract available. PMID 31422126